CLINICAL TRIAL: NCT00470366
Title: Phase II Trial of Paclitaxel, Ifosfamide, and Cisplatin in Previously Untreated Intermediate and Poor Risk Germ Cell Tumor Patients
Brief Title: Combination Chemotherapy and Pegfilgrastim in Treating Patients With Previously Untreated Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-044; MSKCC-07044
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2017-10-24 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2016-06

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Ovarian Cancer; Teratoma; Testicular Germ Cell Tumor
Keywords: stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and seminoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma; testicular embryonal carcinoma and seminoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma; testicular seminoma; testicular yolk sac tumor and teratoma with seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor; stage I malignant testicular germ cell tumor; adult central nervous system germ cell tumor; ovarian choriocarcinoma; ovarian dysgerminoma; ovarian embryonal carcinoma; ovarian yolk sac tumor; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian polyembryoma; ovarian mixed germ cell tumor; stage IV ovarian germ cell tumor; stage IV extragonadal seminoma; stage I extragonadal non-seminomatous germ cell tumor; stage II extragonadal non-seminomatous germ cell tumor; stage III extragonadal non-seminomatous germ cell tumor; stage IV extragonadal non-seminomatous germ cell tumor; adult teratoma; testicular immature teratoma; testicular mature teratoma; stage IA ovarian germ cell tumor; stage IB ovarian germ cell tumor; stage IC ovarian germ cell tumor; stage IIA ovarian germ cell tumor; stage IIB ovarian germ cell tumor; stage IIC ovarian germ cell tumor; stage IIIA ovarian germ cell tumor; stage IIIB ovarian germ cell tumor; stage IIIC ovarian germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Carcinoma, Embryonal; Seminoma; Endodermal Sinus Tumor; Dysgerminoma | interventions — pegfilgrastim; Cisplatin; Ifosfamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel, Ifosfamide, and Cisplatin (Experimental): -Paclitaxel is administered first, 120 mg/m2 on days 1 and 2 every three weeks for four cycles. Cisplatin is administered at 20 mg/m2 over approximately 30 minutes daily for five days every three weeks for four courses. -The ifosfamide is given last with 1200 mg/m2 daily for five days every three weeks for four cycles.
  Interventions: Biological: pegfilgrastim; Drug: cisplatin; Drug: ifosfamide; Drug: paclitaxel

INTERVENTIONS:
Biological: pegfilgrastim
Drug: cisplatin
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, ifosfamide, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy.

PURPOSE: This phase II trial is studying the side effects and how well giving combination chemotherapy together with pegfilgrastim works in treating patients with previously untreated germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of chemotherapy comprising paclitaxel, ifosfamide, and cisplatin in combination with pegfilgrastim in patients with previously untreated intermediate- or poor-risk germ cell tumors.
* Determine the safety of this regimen in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 120-180 minutes on days 1 and 2, cisplatin IV over 30 minutes and ifosfamide IV over 120 minutes on days 1-5, and pegfilgrastim subcutaneously on day 6. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Some patients may required surgery after chemotherapy and, if viable non-teratomatous germ cell tumor is found in the surgical specimen and there is no interval disease progression, these patients may receive 1-2 more courses of chemotherapy after surgery.

After completion of study treatment, patients are followed up at 28 days and then every 2 months for up to 1 year.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed germ cell tumor meeting 1 of the following criteria:

  * Poor risk, defined by any of the following:

    * Testis or retroperitoneal primary site nonseminoma histology without visceral metastases but with "poor-risk" markers, defined by any of the following:

      * Pretreatment serum lactate dehydrogenase (LDH) > 10 times upper limit of normal (ULN)
      * Pretreatment serum human chorionic gonadotropin (HCG) > 50,000 IU/L
      * Pretreatment serum alpha fetoprotein (AFP) > 10,000 ng/mL
    * Testis or retroperitoneal primary site nonseminoma histology with one or more nonpulmonary visceral metastases, including any of the following (regardless of serum tumor marker values):

      * Bone metastases
      * Brain metastases
      * Hepatic metastases
      * Any nonpulmonary metastases (i.e., skin, spleen)
    * Mediastinal primary site nonseminoma histology regardless of serum tumor marker levels or presence/absence of visceral metastases
  * Modified intermediate risk, defined by any of the following:

    * Testis or retroperitoneal primary site nonseminoma histology with no nonpulmonary visceral metastases, and with any of the following serum marker values:

      * Pretreatment serum LDH 3.0-10 times ULN
      * Pretreatment serum HCG 5,000-50,000 IU/L
      * Pretreatment serum AFP 1,000-10,000 ng/mL
    * Seminoma histology with one or more nonpulmonary visceral metastases, including any of the following (regardless of serum tumor marker values or primary site):

      * Bone metastases
      * Brain metastases
      * Hepatic metastases
      * Any nonpulmonary visceral metastases (i.e., skin, spleen)
* Previously untreated disease
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine normal or creatinine clearance > 50 mL/min (unless renal dysfunction is due to tumor obstructing the ureters)
* AST and ALT ≤ 3 times ULN
* Bilirubin ≤ 2.0 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent malignancy except for nonmelanoma skin cancer
* No known HIV positivity
* No active infections

PRIOR CONCURRENT THERAPY:

* Recovered from prior surgery
* More than 30 days since prior radiotherapy and recovered (unless evidence of progressive disease has been documented)
* No prior chemotherapy
* No other concurrent cytotoxic therapy
* Concurrent radiotherapy and surgery allowed for treatment of brain metastases

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert J. Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 03/27/2007 Protocol Closed to Accrual 8/13/2013 Primary Completion Date 06-13-2016 Recruitment Location is the medical clinic
Groups:
- Paclitaxel, Ifosfamide, and Cisplatin: -Paclitaxel is administered first, 120 mg/m2 on days 1 and 2 every three weeks for four cycles. Cisplatin is administered at 20 mg/m2 over approximately 30 minutes daily for five days every three weeks for four courses. -The ifosfamide is given last with 1200 mg/m2 daily for five days every three weeks for four cycles.
  pegfilgrastim
  cisplatin
  ifosfamide
  paclitaxel
Period: Overall Study
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
Started | 60
Completed | 56
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Poor compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 28 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 51
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
Number analyzed (Participants) | 56
Participants
  Complete Response | 38
  PR-Negative | 7
  Incomplete Response | 11

2. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 8 years
Measure: Median (Full Range); unit: years
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
Number analyzed (Participants) | 60
years | 4.4 [1 to 7.6]

3. Secondary Outcome: Percentage of Participants With Progression Free Survival
Description: Progression Free Survival at 3 years. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
Number analyzed (Participants) | 60
percentage of patients | 72 [61 to 84]

4. Secondary Outcome: Number of Patients With Treatment Related Toxicity
Description: Toxicity evaluated and graded according to the National Cancer Institute, Version 3.0
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
Number analyzed (Participants) | 60
Participants | 60

ADVERSE EVENTS:
Time Frame: Day 1, 8 and 15 during each treatment cycle (1 cycle = 21 days). Follow up evaluation will be assessed after 28 days off study as often as every 4-8 weeks for the first year for patients who complete study or withdraw for reason other than progression of disease. For patients who come off study for disease progression, follow-up as often as every 8 weeks for the first year.
Arm/Group | Paclitaxel, Ifosfamide, and Cisplatin
All-Cause Mortality (participants affected / at risk) | 5/60
Serious Adverse Events (participants affected / at risk) | 34/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel, Ifosfamide, and Cisplatin (N=60)
Allergy/Immunology, other (Immune system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1
Cardiac General, other (Cardiac disorders) | 2
Chyle or lymph leakage (Vascular disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine (Investigations) | 3
Cystitis (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 9
Fever (in the absence of neutropenia) (General disorders) | 1
Hematoma (Vascular disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Hemorrhage, Duodenum (Gastrointestinal disorders) | 1
Hemorrhage, Esophagus (Gastrointestinal disorders) | 1
Hypotension (Vascular disorders) | 5
Infection w/ Gr 3/4 Neut, Kidney (Infections and infestations) | 1
Leukocytes (Investigations) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Neutrophils/granulocytes (Investigations) | 10
Obstruction, GU - Ureter (Renal and urinary disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Chest/thorax NOS (General disorders) | 2
Pain - Throat/pharynx/larynx (General disorders) | 3
Platelets (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombosis/embolism (Vascular disorders) | 4
Vomiting (Gastrointestinal disorders) | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel, Ifosfamide, and Cisplatin (N=60)
Nausea (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 17
Hemoglobin (Blood and lymphatic system disorders) | 15
Leukocytes (Investigations) | 13
Neutrophils/granulocytes (Investigations) | 13
Platelets (Investigations) | 13
ALT (Investigations) | 11
Neuropathy: sensory (Nervous system disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 10
AST (Investigations) | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Alkaline phosphatase (Investigations) | 9
Vomiting (Gastrointestinal disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8
Lymphopenia (Investigations) | 7
Tinnitus (Ear and labyrinth disorders) | 7
Hyperbilirubinemia (Investigations) | 6
Diarrhea (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
INR (Investigations) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 5
Amylase (Investigations) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 4
Mucositis - oral cavity (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes